CLINICAL TRIAL: NCT06835725
Title: PHASE II RANDOMIZED TRIAL OF 2- VS 5-FRACTION PROSTATE STEREOTACTIC ABLATIVE RADIOTHERAPY
Brief Title: Phase II Randomized Trial of 2 Versus 5 Fraction Prostate Stereotactic Ablative Radiotherapy for Intermediate Risk Prostate Cancer
Acronym: ADAPT-25
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00030-07; FAS-02207 (Other Grant/Funding Number: BC Cancer Foundation)
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-02

CONDITIONS: Prostate CA
Keywords: stereotactic radiotherapy; SBRT; SABR
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: randomized phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-Fraction Prostate SABR (Experimental): 27Gy delivered to the prostate gland (CTV)in 2 fractions over 2 weeks
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)
- 5-fraction prostate SABR (Active Comparator): 40Gy delivered to the prostate gland (CTV) in 5 fractions over 2 weeks.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — prostate stereotactic ablative radiotherapy
  Other Names: SABR

SUMMARY:
Prostate cancer is a common cancer, and a significant cause of cancer death in men. There are many potentially curative treatment options for prostate cancers that have not spread. A relatively recent option is called prostate stereotactic ablative radiotherapy (SABR). SABR is a form of external beam radiotherapy, where patients receive a small number (5-7) of treatments (also called fractions) of radiation delivered in a highly accurate and precise fashion. Standard prostate SABR is generally given in 5 fractions and has been shown to be at least as effective as conventional external beam radiotherapy. Disease control with SABR appears excellent, and it compares favorably to surgery in terms of side effects and quality of life.

In theory, reducing the number of fractions from 5 to 2 may improve disease control and reduce side effects, in addition to providing added convenience for patients. Small studies suggest prostate SABR in 2 fractions may be highly effective and well tolerated. However, there is little available data comparing 2 and 5 fraction SABR head to head to tell us which is superior.

Two fraction SABR involves delivery of 2 large dose fractions of radiotherapy which could result in significant side effects if proper precautions are not taken. The use of continuous tracking of the prostate gland position during treatment delivery reduces the risk of missing the prostate or overdosing organs near by. Such tracking has been shown to reduce bladder side effects. Also, the use of a rectal spacer placed between the prostate and rectum has been shown to reduce bowel side effects. Also, advanced artificial intelligence (AI)-directed computer applications could potentially improve the targeting of radiation during each treatment.

The ADAPT-2 study is a randomized phase II trial comparing standard 5-fraction SABR with an experimental 2-fraction approach in men with intermediate risk prostate cancer. All treatment, whether 5 or 2-fractions, will use continuous prostate tracking (also called triggered imaging) and a rectal spacer (called Space OAR Hydrogel) to minimize side effects. The trial will also evaluate the potential of a new AI-guided dose guidance application to see if it can improve current methods of targeting SABR each day. This aspect of the study will be offline; that is, the AI application will not be used to actually target treatment for the trial patients. Rather, daily targeting of SABR will use standard conventional means, and the AI application will be studied in a simulated fashion to determine it is useful and can be incorporated into workflow.

The main goal of the ADAPT-25 study is to compare the long-term side effects and quality of life between 5- and 2-fraction prostate SABR. Secondary goals will be to compare the long-term disease control between 5-and 2-fraction prostate SABR, and to evaluate whether a novel AI-directed dose guidance application can be used to better target SABR by reducing doses to neighboring organs, and whether it can be easily fit into prostate SABR workflow.

DETAILED DESCRIPTION:
Purpose:

To compare the late toxicity, quality of life (QOL) and biochemical disease control between prostate stereotactic ablative radiotherapy (SABR) delivered in 2- and 5-fractions for the treatment of intermediate risk prostate cancer. A secondary exploratory analysis is to evaluate, in an offline fashion, the potential utility and feasability of incorporating a novel artificial intelligence-driven dose guidance/adaptive positioning algothim into the image-guidance workflow process for prostate SABR.

Background:

In recent years prostate SABR has emerged as a standard treatment option for low and intermediate risk prostate cancer. Prostate SABR is a precise an accurate form of external beam radiotheapy, typically delivered in 5-7 fractions. The most common dose-fractionation for prostate SABR involves 40Gy to the prostate gland in 5 fractions over 2 weeks.

Multiple randomized trials have established the non-inferiority of prostate SABR in 5-7 fractions compared to conventinal or moderately hypofractionated radiotherapy. In the setting of HDR brachytherapy, 27Gy delivered in 2 fractions is highly convenient and is associated with very high rates of disease control with low toxicity. Two-fraction prostate SABR has been studied in a number of single arm studies, with enouraging results. Cross-study comparison of 2- and 5-fraction SABR suggests the two-fraction regimen may have less bowel and sexual side effects with compariable disease control. Currrently, randomized head-to-head compariosn betweeen 2- and 5-fraction prostate SABR is limited, so it is unknown how the two compare with regard to toxicity, QOL and disease control. Two-fraction SABR is certainly desirable given the potential for improved patient convenience and reduced resource utilization compared to the 5-fraction regimen, and the fact that SABR is less invasive than HDR brachytherapy.

Because of the large dose per fracton of 2-fraction SABR, techniques to minimize toxicity risks are desirable. In this regard, a rectal spacer such as Space OAR Hydrogel is associated with improved toxicity and QOL with prostate radiotherapy and is standard at our institution. Also, real-time prostate tracking is associated with reduced urinary toxicity. Incorporation of these technologies can minimize the risk of treamtent, whether delivered in 2- or 5-fractions.

Also, theortically, improvements in image-guidance that allow for real time dose assessment and adaptive positioning could be used to improve treatment delivery and reduce toxicity. LIMBUS/RADFORMATION have developed a novel AI-driven dose-guidance application that allows for real time assessment of organ at risk and target dose at the time of cone-beam CT at the treatment unit, and can also provide data for adaptive positioning to optimize dose delivery. Study of this technology in the offline setting can provide insight as to the potential utility of the application and how to fit it into prostate SABR worklow, provding the first step before the future online testing of the product.

Given the data above, the present protocol proposes a randomized phase II trial of prostate SABR with the use of a rectal spacer and real-time tracking, comparing 27Gy in 2 weekly fractions and 40Gy in 5 fractions given every other day over 2 weeks, with offline evaluation of an AI-driven dose guidance/adaptive positioning application.

Trial Design:

100 patients with intermediate risk prostate cancer will be randomized 1:1 to prostate SABR with a dose-fractionation of either, (A) 27Gy in 2 fractions over 2 weeks, or (B) 40Gy in 5 fractions over 2 weeks. All patietns will undego fiducial marker and rectal spacer insertion prior to treatment. CT simulation and MR imaging are necessary for treatment planning. Treatments will proceed using a VMAT-based planning and delivery technique. Online image-guidance will involve CBCT and prostate tracking with triggered imaging. The RADFORMATION/LIMBUS dose guidance/adaptive positioning will be applied offline for data collection purposes only.

Patients will be assessed at baseline and in followup with regard to PSA, testosterone, provider-reported toxcity (RTOG and CTCAEv5 scales), and patient-reported outcomes (EPIC-26 bowel/bladder/sexual domains). Subject follow-up will contiue for 5 years after completion of SABR.

Six months of androgen-deprivation therapy is permitted at the discretion of the treating physican. Participants may not be on cytoxic chemotherapy while on SABR. For example, subjects taking methotrexate for benign disease, such as rheumatoid arthritis, must stop the medication during radiotherapy.

Schedule of Assessements:

* Complete history and physical exam including digital rectal examination (DRE), along with assessment of ECOG performance status must be performed within the 16 weeks preceding the start of radiotherapy.
* Pathologic confirmation of adenocarcinoma of the prostate within 18 months of randomization is required.
* CT abdomen/pelvis within 6 months of randomization (may be omitted for NCCN low risk participants).
* Bone scan within 6 months of randomization (may be omitted for NCCN low risk participants).
* Estimation of prostate volume within 6 months of randomization - this can be estimated by imaging (CT, MRI, US) or by DRE. Prostate volume must be estimated to be less than 100cc.
* PSA and testosterone measured within 90 days prior to randomization.
* Baseline symptom assessment using the CTCAE version 5.0 and RTOG/SOMA bladder and bowel toxicity scoring should be performed within the 16 weeks preceding start of radiotherapy
* Baseline participant questionnaires, including the International Prostate Symptom Score (IPSS) and the Expanded Prostate Index Composite-26 Short form (EPIC-26) should be performed within the 16 weeks preceding start of radiotherapy.

Formal Stopping Rules:

The primary objective of this study is to determine and compare the late grade 2+ toxicity at 4 years between arms, thus accrual will continue until the total sample of 100 participants is obtained. However, the trial may be suspended/terminated under certain events as outlined below:

If there are 3 or more major complications (grade 3 or higher toxicity) in the first 11 participants in the 2-fraction arm, or 7 or more during accrual of the 2-fraction arm, then the lower limit of the 95% confidence interval of the true complication rate would be at least 6%, assuming a binomial distribution, and strong consideration will be given to suspend or terminate the trial. In this regard, the Data Monitoring and Safety Committee would review the toxicities and make a recommendation on suspension or termination of the trial.

Endpoints for evaluation:

Primary endpoint: Freedom from grade 2 or higher late toxicity (combined GU + GI) at four years post-treatment.

Secondary endpoints:

i. Freedom from grade 2 or higher acute toxicity (combined GU + GI) at 6 months post-treatment.

ii. Percentage of participants in each arm with a minimally-important change in EPIC-26 bladder, bowel and sexual QOL domains at 6 months (early) and 4 years (late).

iii. Percentage of participants in each arm with moderate to severe urinary symptoms (IPSS≥8) at 6 months (early) and 4 years (late).

iv. 5-year biochemical control in each arm evaluated using the Phoenix (nadir + 2) definition of biochemical failure.

v. Mean dose reduction to the organs at risk (OARs) using RADFORMATION dose-guided adaptive positioning, offline.

vi. Percentage of fractions in which the parallel, offline use of the RADFORMATION dose-guidance algorithm could be utilized without exceeding the time constraints of a standard treatment slot.

Sample Size Calculation:

The study will use a screening-type phase II design. With α of 0.2 the sample size of 100 subjects randomized 1:1 to each arm provides 80% power to detect a 20% difference in cumulative late grade 2 toxicity (combined GI + GU) at 4 years.

Planned Study Period:

Based on the rate of enrollment on the BC Cancer Prostate SABR registry and the previous ASSERT trial, the estimated accrual period is 3 years. Subsequently, 5 years of follow-up is required after the last participant is randomized. Therefore, the total study duration is estimated at 8 years after commencement of accrual.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 or older.

  * Able to provide informed consent.
  * ECOG performance status 0 - 2.
  * Fit for all protocol treatment and follow-up.
  * Life Expectancy > 5 years.
  * Histologically confirmed adenocarcinoma of the prostate, NCCN low or intermediate risk, with biopsy performed within the last 18 months:

Low risk = cT1-T2a,Gleason ≤ 6, and PSA < 10ng/mL. Intermediate risk = at least one of: cT2b/T2c, PSA 10-20ng/mL, or Gleason 7, but not high risk.

* 6 months of Androgen Deprivation Therapy (ADT) is permitted for those with NCCN unfavorable intermediate risk disease (aka high-tier intermediate risk disease), defined as intermediate risk disease with one or more of: two or three intermediate risk features, Gleason 4+3, or ≥50% biopsy cores positive.
* For those with NCCN unfavorable intermediate risk disease, it is permitted for ADT to have been initiated prior to study enrollment provided it is possible for radiotherapy to be completed before completion of 6 months of ADT.
* Prostate volume <100cc based on imaging or digital rectal examination.
* PSA within 90 days prior to registration. If ADT is started before registration, then the PSA must have been done no more than 90 day prior to the date of the first ADT injection.
* CT abdomen and pelvis within the 6 months prior to registration (may be omitted for NCCN low risk participants). If particpant started on ADT prior to registration, CT should be done before first ADT injection.
* Bone scan within the 6 months prior to of registration (may be omitted for NCCN low risk participants). If particpant started on ADT prior to registration, bone scan should be done before first ADT injection.
* Must be appropriate for and willing to undergo implantation of prostate fiducial markers and Space OAR Hydrogel.

Exclusion Criteria:

Clinical stage cT3 or greater. Gleason score 8 or greater. PSA > 20ng/mL or greater. NCCN high or very high risk. Pelvic nodal metastases. Distant metastases. Previous malignancy within the last 5 years except basal or squamous cell carcinomas of the skin.

Previous pelvic radiotherapy. Any prior active local treatment for prostate cancer. Participants previously on active surveillance are eligible if they continue to meet all other eligibility criteria.

Unilateral or Bilateral hip prostheses. Medical conditions likely to make radiotherapy inadvisable (e.g., inflammatory bowel disease).

Medical condition that would make implantation of fiducial markers or hydrogel rectal spacer unsafe, in the opinion of the treating physician (e.g., pelvic or prostate abscess).

Medical condition or implant that prohibits MRI (e.g. pacemaker) Trans-urethral resection of the prostate (TURP), GreenLight Laser or Holmium Laser Prostate procedure within 6 months of radiotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients must have a prostate gland
Enrollment: 100 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2032-04-30 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from grade 2 or higher toxicity | At Four years after treatment
  proportion of patients without grade 2 or higher GU or GI toxicity

SECONDARY OUTCOMES:
Freedom from grade 2 or higher acute toxicity | 6 months post-treatment
  Proportion of patients free of grade 2 or higher acute GI or GU toxicity
quality of life | At Four years after treatment
  proportion of patients in each arm with a MID in EPIC-26 quality of life
5-year biochemical recurrence-free survivial | Five years
  proportion of patients free of biochemical recurrence
feasibility of AI-dose guidance | estimate 3 years (when all patients accrued and treated)
  Percentage of fractions that AI application could be run within treatment time slot, and the offline organ at risk dose reduction by using the adaptive positioning aspect of the application

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Alexander, Principal Investigator — BC Cancer; Winkle Kwan, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer Radiation Oncology, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Depends on BC Cancer institutional regulations